CLINICAL TRIAL: NCT01444768
Title: Prospective Evaluation of Computerized Physician Order Entry in the Emergency Department
Acronym: CPOE
Status: Withdrawn | Type: Observational
Sponsor: Beth Israel Deaconess Medical Center (Other)
Responsible Party: Principal Investigator, Steven Horng, MD, Instructor in Emergency Medicine, Beth Israel Deaconess Medical Center
Other Study IDs: 2011P000308
Record Dates: First submitted 2011-09-29; First posted 2011-10-03 (Estimated); Last update posted 2017-04-05 (Actual); Status verified 2017-04

CONDITIONS: Operational Metrics of the Emergency Department
Keywords: Alert Systems, Medication; Computerized Physician Order Entry System; CPOE; Medication Alert Systems; Medical Order Entry Systems
MeSH Terms: interventions — Medical Order Entry Systems

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Other: Computerized Physician Order Entry — Computer ordering system allowing emergency department physicians to order medications, laboratory tests, radiology studies, and nursing interventions

SUMMARY:
This study will evaluate various performance metrics of emergency department operations after the implementation of computerized physician order entry in an academic emergency department.

DETAILED DESCRIPTION:
The study will be a prospective before-after study comparing various operational and performance metrics before and after the implementation of a computerized physician order entry system in the emergency department.

The investigators will collect 6 month before, 6 month after of data along with a 2-4 week washout period. The investigators will also administer a computerized physician order entry survey after the study is completed. This confidential survey will be emailed to all ED nurses, residents, and attendings using RedCap. Consent will be implied if they choose to participate.

ELIGIBILITY:
Inclusion Criteria:

* All consecutive adult patients (Age >=18) presenting to the Emergency Department during the study period will be included in the study.

Exclusion Criteria:

* Patients who eloped, left without being seen, or signed out against medical advice will be excluded.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: All patients who are registered in the emergency department > 18 years of age who do not elope, left without being seen, or leave AMA.
Sampling Method: Non-Probability Sample
Enrollment: 0 (Actual)
Dates: Start 2012-03; Primary Completion 2012-12 (Estimated); Study Completion 2013-12 (Estimated)

PRIMARY OUTCOMES:
Time to Antibiotics | 6 months
  Primary outcome measure is time to antibiotics. This is defined as the time patients are registered to the time they receive their first antibiotics for patients with an ED diagnosis of pneumonia.

SECONDARY OUTCOMES:
Emergency Department Length of Stay | 6 months
  Secondary outcome measure is length of stay defined as the time from patient registration to time the patients leave the emergency department.
Lab turnaround time | 6 months
  Lab turnaround time is defined as the time it takes from when the sample is collected to when the results are entered.
Resource Utilization | 6 months
  Resource utilization defined as the number of CBC, Chem7, and troponin tests ordered.

CONTACTS AND LOCATIONS:
Overall Officials: Steven Horng, MD, Principal Investigator — Beth Israel Deaconess Medical Center
Locations (1):
- Beth Israel Deaconess Medical Center, Boston, Massachusetts, United States